CLINICAL TRIAL: NCT01769235
Title: A Multicenter, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Taro Pharmaceutical Inc.'s Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5% to the Reference Listed Acanya® (Clindamycin Phosphate and Benzoyl Peroxide)Gel, 1.2%/2.5% and Both Active Treatments to a Vehicle Control in the Treatment of Acne Vulgaris
Brief Title: Study Comparing Clindamycin Phosphate and Benzoyl Peroxide Gel to Acanya® Gel and Both to a Vehicle Control in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLBG 1210
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Clindamycin Phosphate and Benzoyl Peroxide Gel; Acanya® Gel
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5% (Experimental): Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5% (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5%
- Acanya® Gel, 1.2%/2.5% (Active Comparator): Acanya® (Clindamycin Phosphate and Benzoyl Peroxide) Gel, 1.2%/2.5% (Dow Pharmaceutical Sciences, Inc., marketed by Valeant Pharmaceuticals North America LLC)
  Interventions: Drug: Acanya® Gel, 1.2%/2.5%
- Vehicle of test product (Placebo Comparator): Vehicle of test product (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Vehicle of test product

INTERVENTIONS:
Drug: Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5% — Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5% (Taro Pharmaceuticals Inc.)applied at approximately the same time once daily for 84 days (12 weeks).
  Arms: Clindamycin Phosphate and Benzoyl Peroxide Gel, 1.2%/2.5%
Drug: Acanya® Gel, 1.2%/2.5% — Acanya® (Clindamycin Phosphate and Benzoyl Peroxide) Gel, 1.2%/2.5% (Dow Pharmaceutical Sciences, Inc., marketed by Valeant Pharmaceuticals North America LLC)applied at approximately the same time once daily for 84 days (12 weeks).
  Arms: Acanya® Gel, 1.2%/2.5%
Drug: Vehicle of test product — Vehicle of test product (Taro Pharmaceuticals Inc.)applied at approximately the same time once daily for 84 days (12 weeks).
  Arms: Vehicle of test product

SUMMARY:
The objective of this study is to compare the safety and efficacy profiles of Taro Pharmaceutical Inc.'s Clindamycin Phosphate and Benzoyl Peroxide Gel 1.2%/2.5% to Acanya® (Clindamycin Phosphate and Benzoyl Peroxide) Gel, 1.2%/2.5% and to demonstrate the superior efficacy of the two active formulations over that of the vehicle in the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the study.
* Be 12 to 40 years of age, inclusive. A subject may be of either sex and any race/ethnicity.
* Have a clinical diagnosis of facial acne vulgaris with 25 or greater non-inflammatory lesions and 20 or greater inflammatory lesions and no more than 2 nodulocystic lesions.
* Have a baseline Investigator's Global Assessment of acne severity grade of 2, 3 or 4 on a severity scale of 0 to 4.
* Be willing and able to understand and comply with the requirements of the study, apply the study medication as instructed, refrain from use of all other topical acne medication and topical antibiotics during the 12-week treatment period, return for the required treatment period visits, comply with therapy prohibitions, and able to complete the study.
* Be in general good health and free from any clinically significant disease, other than acne vulgaris, that might interfere with the study evaluations.
* Female subjects of childbearing potential must have a negative urine pregnancy test amd must be willing to use a medically accepted method of contraception during the study.

Exclusion Criteria:

* Presence of more than 2 facial nodulocystic lesions (i.e., nodules and cysts).
* Current diagnosis of acne conglobata, acne fulminans, or secondary acne.
* Presence of active cystic acne, or polycystic ovarian syndrome.
* History or presence of Crohn's disease, ulcerative colitis, regional enteritis, or antibiotic-associated colitis.
* Presence of any other facial skin condition that might interfere with acne vulgaris diagnosis and/or assessment.
* Excessive facial hair that would interfere with diagnosis or assessment of acne vulgaris.
* History of unresponsiveness to topical clindamycin phosphate and/or benzoyl peroxide therapy.
* Start or change of dose of estrogens or hormonal treatment 3 months prior to baseline or throughout the study.
* Use of medicated make-up throughout the study and significant change in the use of consumer products within 30 days of study entry and throughout the study.
* Use of any of the following treatments more recently than the indicated washout period prior to visit 1/day 1; need or intent to continue to use any of the following treatments during the study: oral retinoids or therapeutic Vitamin A supplements of greater than 10,000 units/day; systemic steroids; systemic antibiotics; systemic treatment for acne vulgaris ; systemic anti-inflammatory or immunosuppressive agents (NSAID use is allowed on an as-needed basis but for no more than 7 days of consecutive use, low dose aspirin is allowed if on a stable dose for at least 30 days); Spironolactone; use on the face of cryodestruction or chemodestruction, dermabrasion, photodynamic therapy, acne surgery, intralesional steroids, x-ray therapy; topical retinoids; topical steroids; topical anti-acne medications; topical anti-inflammatory agents; topical antibiotics; medicated cleansers; use of tanning booths, sun lamps, sunbathing or excessive exposure to the sun; antipruritics, including antihistamines.
* History of hypersensitivity or allergy to clindamycin phosphate, benzoyl peroxide, and /or any ingredient in the study medication.
* Females who are pregnant, breastfeeding, intending to become pregnant during the study, or who do not agree to use an acceptable form of birth control during the study.
* Consumption of excessive alcohol, abuse of drugs, or a condition that could compromise the subject's ability to comply with study requirements.
* Any clinically significant condition or situation other than acne vulgaris that would interfere with the study evaluations or optimal participation.
* Use of any investigational drugs within 30 days prior to visit 1/day 1.
* Participation in any other clinical study in the 30 days prior to signing the informed consent form.
* Previous participation in this study.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1215 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Mean percent change in inflammatory lesion counts. | 12 weeks
  Mean percent change from baseline to week 12 in the inflammatory (papules and pustules) lesion counts.
Mean percent change in non-inflammatory lesion counts. | 12 weeks
  Mean percent change from baseline to week 12 in the non-inflammatory (open and closed comedones) lesion counts.

SECONDARY OUTCOMES:
Clinical response of "success". | 12 weeks
  The proportion of subjects at week 12 with a clinical response of "success" is defined as an Investigators Global Assessment score that is at least 2 grades less than the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Symbio CRO, Study Chair — http://symbioresearch.com/